CLINICAL TRIAL: NCT01999803
Title: A Phase I, Randomised, Double-blind, Placebo-controlled Study in Patients With Amyotrophic Lateral Sclerosis to Further Assess the Safety and Tolerability of Intracerebroventricular Administration of sNN0029 Infusion Solution
Brief Title: A Safety Study of sNN0029 Administration Via Intracerebroventricular Route to Patients With ALS
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Issues with development and supply of infusion system for delivery of IMP. Lack of favorable benefit risk ratio in sNN0029-003 study (review of interim data).
Sponsor: Newron Sweden AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: sNN0029-003; 2012-001026-10 (EudraCT Number)
Record Dates: First submitted 2013-11-22; First posted 2013-12-03 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sNN0029 (VEGF) (Experimental): 4 µg/d of sNN0029 administered by continuous intracerebral infusion during12 weeks
  Interventions: Drug: sNN0029
- Placebo (Placebo Comparator): Placebo administered by continuous intracerebral infusion during12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: sNN0029
  Other Names: telbermin, rhVEGF165
  Arms: sNN0029 (VEGF)
Drug: Placebo
  Other Names: Artificial CSF
  Arms: Placebo

SUMMARY:
This is a phase I, multicentre randomised, double-blind, placebo-controlled trial to assess the safety and tolerability of continuous i.c.v. administration of sNN0029 infusion solution at a dose of 4µg/day in patients with Amyotrophic Lateral Sclerosis (ALS).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of ALS classified as definite, or probable with or without additional laboratory evidence, according to the revised World Federation of Neurology (WFN) El Escorial criteria.
* If patients are being treated with riluzole, they must have been on a stable dose for at least the past 30 days prior to screening.
* The patient is, in the opinion of the investigator, medically fit to undergo the surgery required for stereotactic implantation of the catheter and infusion pump.

Exclusion Criteria:

1. Impaired respiratory function judged to pose a risk to the patient during anaesthesia for the device implantation.
2. Hypertension defined as blood pressure >160 mmHg systolic or >90 mmHg diastolic.
3. Values for coagulation parameters including platelet count, normalised prothrombin complex (PK-INR), activated partial thromboplastin time (APTT) outside normal ranges.
4. Ophthalmological examination (fundus photography, visual acuity and perimetry) with any clinically significant findings that imply safety concerns for this study.
5. Diagnosis of diabetes mellitus.
6. History of structural brain disease other than ALS, including tumours and hyperplasia.
7. An MRI of the brain and cervical spine, and an Magnetic Resonance Angiography (MRA) of the brain with findings of tumours or potential sources of pathological bleedings, or abnormality that may interfere with the assessments of safety or efficacy or that would, in the judgment of the investigator, represent a surgical risk to the patient. If an MRI and/or MRA has been performed within 1 month prior to screening, the results from that examination can be used.
8. Any disorder that precludes a surgical procedure (e.g., signs of sepsis or inadequately treated infection), alters wound healing (e.g., including bleeding disorders), or renders chronic i.c.v. delivery or device implants medically unsuitable.
9. Presence of risk for increased or uncontrolled bleeding and/or risk of bleeding that cannot be not managed optimally due to:

   i. anatomical factors at or near the implant site (e.g., vascular abnormalities, neoplasms, or other abnormalities), ii. underlying disorders of the coagulation cascade, platelet function, or platelet count (e.g., haemophilia, Von Willebrand's disease, liver disease, or other medical conditions) iii. administration of any antiplatelet or anticoagulant medication in the preoperative period
10. A personal history of thromboembolic disease. A family history of thromboembolic disease will prompt a laboratory assessment to exclude hereditary liability before the patient is declared eligible.
11. Presence of additional risk factors for thromboembolism such as obesity (BMI > 35) or use of oestrogens including combined contraceptive pills.
12. Presence of an implanted shunt for the drainage of CSF or an implanted Central Nervous System (CNS) catheter.
13. Clinically significant abnormalities in haematology or clinical chemistry parameters as assessed by the investigator.
14. Serological evidence of Hepatitis B virus (HBV), Hepatitis C virus (HCV) or Human immunodeficiency virus (HIV)
15. Ongoing medical condition that according to the investigator would interfere with the conduct and assessments in the study. Examples are medical disability (e.g., severe degenerative arthritis, compromised nutritional state, peripheral neuropathy) that would interfere with the assessment of safety and efficacy of investigational product or device performance, or would compromise the ability of the patient to undergo study procedures (e.g., MRI), or to give informed consent.
16. Participation in another clinical trial with an investigational drug or device within 3 months prior to screening visit.
17. For women only: pregnant, breast feeding and/or for fecund women unwillingness to use adequate contraception during the trial such as:

    * Established use of oral, injected or implanted hormonal methods of contraception that do NOT contain oestrogens.
    * Placement of an intrauterine device.
    * Barrier methods of contraception: Condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-09; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events (AEs) | 12 weeks
  The safety and tolerability of i.c.v. administration of sNN0029 infusion solution at a dose of 4 µg/day delivered via a Medtronic SynchroMed® II Infusion System will be evaluated by comparing tabulated number of events over 12 weeks by body system, preferred term and by severity and relationship to study medication/device. Serious Adverse Events/Serious Adverse Device Events will also be presented in separate tabulations.

SECONDARY OUTCOMES:
VEGF165 levels in Cerebrospinal Fluid (CSF) | 12 weeks
  Levels of the active ingredient of sNN0029 infusion solution (VEGF165) in CSF will be summarised using descriptive statistics by time point and treatment.
Medical Device performance | 12 weeks
  Device performance (number of values +/-25% of expected) will be presented by time point and treatment.

OTHER OUTCOMES:
ALS Functional Raring Scale - Revised (ALSFRS-R) | 12 weeks
  ALSFRS-R score (0=worst to 48=best) will be analysed as absolute value and as change from baseline using descriptive statistics by time point and treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Philip VanDamme, Prof, MD, Principal Investigator — University Hospital Leuven, Herestraat 49, B-3000 Leuven, Belgium; Leonard van den Berg, MD, Prof, Principal Investigator — University Medical Center Utrecht, Department of Neurology G03.228, P.O. Box 85500, NL-3508 GA Utrecht, The Netherlands
Locations (2):
- Philip Van Damme, Leuven, Belgium
- Leonard van den Berg, Utrecht, Netherlands